CLINICAL TRIAL: NCT05416229
Title: The QUANTUM Trip Trial - Psilocybin-assisted Therapy for Reducing Alcohol Intake in Patients With Alcohol Use Disorder: A Randomized, Double-blinded, Placebo-controlled Clinical Trial.
Brief Title: Psilocybin-assisted Therapy for Treatment of Alcohol Use Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anders Fink-Jensen, MD, DMSci (Other)
Collaborators: The Neurobiology Research Unit at Copenhagen University Hospital Rigshospitalet (Unknown)
Responsible Party: Sponsor-Investigator, Anders Fink-Jensen, MD, DMSci, Professor, Psychiatric Centre Rigshospitalet
Organization: Psychiatric Centre Rigshospitalet (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSILO4ALCO-TRIAL
Record Dates: First submitted 2022-05-30; First posted 2022-06-13 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Alcohol Use Disorder
Keywords: psilocybin; alcohol dependence; addiction; randomized controlled trial; brain imaging
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Psilocybin; maltodextrin

STUDY DESIGN:
Intervention Model Description: single-centre, randomised, double-blinded, placebo-controlled, 1:1 parallel-group clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin-assisted therapy (Experimental): 45 patients will receive a single administration of 25mg psilocybin given in a protocol of psychological support before, during and after dosing.
  Interventions: Drug: Psilocybin
- Placebo-assisted therapy (Placebo Comparator): 45 patients will receive a single administration of placebo (lactose) given in a protocol of psychological support before, during and after dosing.
  Interventions: Drug: Maltodextrin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin-assisted therapy
  Arms: Psilocybin-assisted therapy
Drug: Maltodextrin — Placebo-assisted therapy
  Arms: Placebo-assisted therapy

SUMMARY:
Note: The trial is only eligible for citizens of Denmark.

The purpose of this project is to assess the treatment efficacy of a single high dose of psilocybin administered within a protocol of psychological support to patients diagnosed with alcohol use disorder (AUD).

DETAILED DESCRIPTION:
To establish efficacy, we will investigate a single dose of psilocybin versus placebo in a randomised, double-blinded, placebo-controlled 12 weeks clinical trial. 90 patients, aged 20-70 years, diagnosed with alcohol use disorder and treatment seeking will be recruited from the community via advertisement and referrals from general practitioners and hospital units. The psilocybin or placebo is administered within a protocol of psychological support before, during and after the dosing. Outcome assessments will be carried out one, four, eight- and 12 weeks post dosing. The primary outcome is reduction in the percentage of heavy drinking days from baseline to follow-up at 12 weeks. Key secondary outcomes include 1) phosphatidyl-ethanol as an objective biomarker for alcohol consumption 2) plasma psilocin, the active metabolite, to establish a possible therapeutic range and 3) the acute subjective drug experience as a possible predictor of treatment outcome. Furthermore, we will investigate the neurobiological underpinnings of the possible treatment effects by use of functional magnetic resonance brain imaging one week post dosing.

ELIGIBILITY:
Inclusion Criteria:

* Bodyweight of 50-110 kg
* AUD according to DSM-5 criteria and alcohol dependence according to ICD-10.
* AUD Identification Test (AUDIT) ≥ 15.
* ≥ 5 heavy drinking days in the past 28 days prior to inclusion.

Exclusion Criteria:

* Current or previously diagnosed with any psychotic disorder or bipolar affective disorder.
* Immediate family member with a diagnosed psychotic disorder.
* History of delirium tremens or alcohol withdrawal seizures.
* History of suicide attempt or present suicidal ideation at screening.
* Withdrawal symptoms at screening (>nine on the Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar) (43).
* Present or former severe neurological disease including trauma with loss of consciousness > 30 min.
* Impaired hepatic function (alanine transaminase >210/135 units/l men/women)
* Cardiovascular disease defined as decompensated heart failure (NYHA class III or IV), unstable angina pectoris, myocardial infarction within the last 12 months or uncontrolled hypertension (systolic blood pressure >165 mmHg, diastolic blood pressure >95 mmHg).
* Present or former abnormal QTc (>450/470 ms men/women).
* Treatment with disulfiram, naltrexone, acamprosate and nalmefene within 28 days of inclusion.
* Treatment with any serotonergic medication or drugs within one month prior inclusion.
* Any oOther active substance use disorders (except nicotine) defined as a Drug Use Disorder Identification Test score >six/two (men/women) and investigator's clinical evaluation.
* Women who are pregnant, breastfeeding, or intend to become pregnant or are not using adequate contraceptive measures considered highly effective (44).
* Unable to speak or understand Danish.
* Any other condition that the clinician estimates can interfere with trial participation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of heavy drinking days | Baseline to week 12
  Heavy drinking is defined as days with five drinks/60 grams of alcohol or more for men, four drinks/48 grams of alcohol or more for women. Data will be collected using the Timeline Followback Method (TLFB) which is a widely used, calendar-based retrospective measure of self-reported use of alcohol. The number of days drinking assessed is 28 days.

SECONDARY OUTCOMES:
Change in total alcohol consumption | Baseline to week 12
  Total grams of alcohol consumed per day as measured by TLFB.
Change in days of abstinence | Baseline to week 12
  Percentage of days without any alcohol consumption as measured by TLFB.
Change in phosphatidyl-ethanol (PEth) | Baseline to week 12
  PEth is formed only in the presence of alcohol and is correlated with the amount of alcohol consumed the past month. PEth concentrations will be measured by peripheral blood test.
Change in Alcohol Use Disorders Identification Test (AUDIT) | Baseline to week 12
  AUDIT is a 10-item questionnaire that measures alcohol use. The score range is 0-40, with higher scores indicating a more problematic use of alcohol.
Change in Penn Alcohol Craving Scale (PACS) score | Baseline to week 12
  PACS is a 40-item questionnaire that measures alcohol craving severity. The score range is 0-30, with higher scores indicating more severe symptoms.
Change in Alcohol Abstinence Self-efficacy Scale (AASE) score | Baseline to week 12
  AASE is a 40-item questionnaire that measures two scales: the temptation to drink and the confidence in the ability to avoid drinking. The score range for each scale is 0-80, with higher score indicating greater temptation or confidence, respectively.
Change in Fagerstrom Test for Nicotine Dependence (FTND) | Baseline to week 12
  FTND is a 6-item questionnaire that measures the quantity of cigarette consumption, the compulsion to use, and dependence. The score range is 0-10, with higher scores indicating a more severe dependence.
Change in Drug Use Disorders Identification Test (DUDIT) | Baseline to week 12
  DUDIT is an 11-item questionnaire that measures drug use. The score range is 0-44, with higher scores indication a more problematic use.
Change in Major Depression Inventory (MDI) | Baseline to week 12
  MDI is a 12-item questionnaire that measures depression severity. The score range is 0-50, with higher scores indicating greater severity.
Change in Short-Form 36 (SF-36) | Baseline to week 12
  SF-36 is a 36-item questionnaire that measures the quality-of-life. The score range is 0-100, with higher scores indicating better health status.
Change in Mindful Attention Awareness Scale (MAAS) | Baseline to week 12
  MAAS is a 15-item scale that measures core characteristic of mindfulness. The score range is 1-6, with higher scores indicating greater mindfulness.
Change in Acceptance and Action Questionnaire (AAQ) | Baseline to week 12
  AAQ is a 7-item questionnaire that measures psychological flexibility. The score range is 7-49, with higher scores indicating lesser flexibility.
Change in NEO-Personality Inventory (NEO-PI= | Baseline to week 12
  The NEO-PI is a 240-item personality instrument that measures the five factors in the Five Factor Model. It consists of 30 eight-item facet scales, 6 for each of the five basic personality factors: Neuroticism (N), Extraversion (E), Openness (O), Agreeableness (A), and Conscientiousness (C), rated by use of a 5-point Likert-type scale ranging from strongly disagree to strongly agree.
Persisting Effects Questionnaire (PEQ) | Week 12
  PEQ is a 143-item scale aiming to assess changes in attitudes, moods, behavior, and spiritual experience
Neuroplasticity and inflammation | Baseline to week 12
  Neuroplasticity and inflammation as measured by mean concentrations of plasma serum brain-derived neurotrophic factor (BDNF) and plasma cytokines, respectively.
Subjective effects of psilocybin: Subjective Drug Intensity (SDI) | 0-6 hours post dosing
  SDI will be regularly assessed asking the patients "how intense is the experience right now" on a 0-10 Likert scale where 0 = not intense at all, 10 = very intense.
Pharmacokinetics- and dynamics of psilocybin | 0 - 6 hours post dosing
  Pharmacokinetics- and dynamics of plasma psilocin, serum BDNF and plasma cytokines, as determined by concentration-time curves of mean plasma concentrations
Subjective effects of psilocybin: Mystical Experience Questionnaire (MEQ) | Completed once the effects are fully subsided or at least 6 hours after dosing
  MEQ is a 30-item questionnaire that measures experiential aspects of psilocybin. The patients are asked to rate the items on a 6-point scale going from 0= none; not at all to 5=extreme; more than ever before in my life and stronger than 4.
Subjective effects of psilocybin: 5-Dimensional Altered State of Consciousness scale (5D-ASC) | Completed once the effects are fully subsided or at least 6 hours after dosing
  5D-ASC is a 94-item questionnaire that measures experiential aspects of psilocybin. The patients are asked to rate the items by placing marks on a horizontal visual analogue scale (100 millimeters in length) going from "no, not more than usual" (on the left) to "yes, very much more than usual" (on the right).
Subjective effects of psilocybin: Ego Dissolution Inventory (EDI) | Completed once the effects are fully subsided or at least 6 hours after dosing
  EDI is a 8-item questionnaire that measures the experiential aspects of psilocybin. The patients are asked to rate the items by placing marks on a horizontal visual analogue scale (100 millimeters in length) going from "no, not more than usual" (on the left) to "yes, very much more than usual" (on the right).
Subjective effects of psilocybin: Emotional Breakthrough Inventory (EBI) | Completed once the effects are fully subsided or at least 6 hours after dosing
  EBI is a 6-item questionnaire that measures the experiential aspects of psilocybin. The patients are asked to rate the items by placing marks on a horizontal visual analogue scale (100 millimeters in length) going from "no, not more than usual" (on the left) to "yes, very much more than usual" (on the right).
Subjective effects of psilocybin: Awe Experience Scale (AWE-S) | Completed once the effects are fully subsided or at least 6 hours after dosing
  AWE-S is a 30-item questionnaire that measures the experiential aspects of psilocybin. The patients are asked to rate the items on a 7-point scale going from 1= Strongly Disagree to 7= Strongly Agree.
Brain imaging | 1 week post dosing
  The blood-oxygen-level-dependent differences between the two treatment arms with respect to resting-state functional connectivity, alcohol vs neutral cue-reactivity within mesocorticolimbic pathways and habitual vs goal-directed activity within corticostriatal pathways

OTHER OUTCOMES:
Role of the Music I | before and after dosing
  We will explore the role of the music in psilocybin-assisted therapy by use of the questionnaires Experience with Music and Geneva Emotional Music Scale
Role of the Music II | week 4
  We will explore the role of the music in psilocybin-assisted therapy by qualitative semi-structured interview
Treatment expectancies | Baseline
  The Stanford Expectations of Treatment Scale is a 6 item a scale that measures positive and negative treatment expectancies using a Likert scale from 1 (strongly disagree) to 7 (strongly agree)
Optional long-term follow-ups | week 26 and week 52
  Patients may consent to post-trial follow-up to explore the long-term effects on drinking outcomes using TLFB adjusted for current or previous treatments since completing the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fink-Jensen, Professor, Principal Investigator — Psychiatric Center Copenhagen, Frederiksberg Hospital
Locations (1):
- Psychiatric Center Copenhagen, Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Jensen ME, Stenbaek DS, Juul TS, Fisher PM, Ekstrom CT, Knudsen GM, Fink-Jensen A. Psilocybin-assisted therapy for reducing alcohol intake in patients with alcohol use disorder: protocol for a randomised, double-blinded, placebo-controlled 12-week clinical trial (The QUANTUM Trip Trial). BMJ Open. 2022 Oct 14;12(10):e066019. doi: 10.1136/bmjopen-2022-066019. PMID 36241352